CLINICAL TRIAL: NCT01016886
Title: A Prospective Study to See if Cardiac Effects of Herceptin Can be Prevented With Standard Heart Medications
Brief Title: Multidisciplinary Approach to Novel Therapies in Cardiology Oncology Research
Acronym: MANTICORE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Organization: AHS Cancer Control Alberta (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 00027 / Ethics 25253
Record Dates: First submitted 2009-11-18; First posted 2009-11-20 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer; Heart Failure
Keywords: trastuzumab; cardiac MRI; beta-blocker; biomarkers; angiotensin converting enzyme inhibitor; cardiotoxicity; HER2 positive
MeSH Terms: conditions — Breast Neoplasms; Heart Failure; Cardiotoxicity | interventions — Perindopril; Bisoprolol

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: perindopril OR bisoprolol OR placebo

INTERVENTIONS:
Drug: perindopril OR bisoprolol OR placebo — perindopril- oral daily titrated does from 2mg up to 8mg
  bisoprolol- oral daily titrated dose from 2.5mg up to 10mg

SUMMARY:
While trastuzumab has been shown to prevent recurrences of breast cancer, some women may also experience damage to their heart muscle (including heart failure) as a result of their treatment. The investigators hope to learn if standard medications used in heart failure can prevent heart damage caused by trastuzumab in women with breast cancer. The investigators would also like to know if there are any ways to detect this damage earlier using magnetic resonance imaging (MRI) and blood tests.

DETAILED DESCRIPTION:
We propose a randomized, placebo-controlled, double-blind study evaluating the efficacy of an ACE-inhibitor (perindopril) or a beta blocker (bisoprolol) for the prevention of LV remodeling among women with early breast cancer scheduled for chemotherapy and one year of trastuzumab. Participants will undergo cardiac MRI at baseline and 3 and 12 months, replacing the usual MUGA, as well as a post-treatment cardiac MRI at 24 months to evaluate long-term effect.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of HER2 positive breast carcinoma
* Eligible to receive trastuzumab
* Age > 18 years
* Able to give informed consent
* No contraindications to MRI

Exclusion Criteria:

* Known contraindication to beta-blocker therapy
* Known contraindication to ACEI therapy
* Current treatment with ACEI or beta blocker for other indication
* History of heart failure, cardiomyopathy or baseline LVEF < 50%

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-09; Primary Completion 2015-09 (Actual); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to determine if conventional heart failure pharmacotherapy can prevent trastuzumab-mediated left ventricular (LV) remodeling among women with HER2+ early breast cancer. | 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ian Paterson, MD FRCPC, Principal Investigator — Alberta Health services
Locations (1):
- University of Alberta/ Cross Cancer Institute, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Haykowsky MJ, Mackey JR, Thompson RB, Jones LW, Paterson DI. Adjuvant trastuzumab induces ventricular remodeling despite aerobic exercise training. Clin Cancer Res. 2009 Aug 1;15(15):4963-7. doi: 10.1158/1078-0432.CCR-09-0628. Epub 2009 Jul 21. PMID 19622583
- [Derived] Pituskin E, Haykowsky M, Mackey JR, Thompson RB, Ezekowitz J, Koshman S, Oudit G, Chow K, Pagano JJ, Paterson I. Rationale and design of the Multidisciplinary Approach to Novel Therapies in Cardiology Oncology Research Trial (MANTICORE 101--Breast): a randomized, placebo-controlled trial to determine if conventional heart failure pharmacotherapy can prevent trastuzumab-mediated left ventricular remodeling among patients with HER2+ early breast cancer using cardiac MRI. BMC Cancer. 2011 Jul 27;11:318. doi: 10.1186/1471-2407-11-318. PMID 21794114